CLINICAL TRIAL: NCT02250976
Title: A Clinical Trial to Evaluate the Pharmacokinetics of the Fixed-dose Combination of Micronized Fenofibrate and Pitavastatin Ca Under Fed Condition in Healthy Male Volunteers
Brief Title: The Pharmacokinetic Study of the Fixed-dose Combination of Micronized Fenofibrate and Pitavastatin Ca
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HL-PIF-103
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Livasupril Cap.160/2mg (Experimental): * Fenofibrate pellet ( as micronized fenofibrate 160mg) and Pitavastatin Ca 2mg
  * once a day
  Interventions: Drug: Livasupril Cap.160/2mg
- Lipilfen cap.160mg, Livaro tab. 2mg (Active Comparator): * Lipilfen cap.160mg : Micronized fenofibrate 160mg , Livaro tab. 2mg : Pitavastatin ca 2mg
  * Coadministariton of Lipilfen cap.160mg and Livaro tab. 2mg, once a day
  Interventions: Drug: Lipilfen cap. 160mg; Drug: Livaro tab. 2mg

INTERVENTIONS:
Drug: Livasupril Cap.160/2mg — Fenofibrate pellet( as micronized fenofibrate 160mg) and Pitavastatin Ca 2mg
  Arms: Livasupril Cap.160/2mg
Drug: Lipilfen cap. 160mg — Micronized fenofibrate 160mg
  Arms: Lipilfen cap.160mg, Livaro tab. 2mg
Drug: Livaro tab. 2mg — Pitavastatin Ca 2mg
  Arms: Lipilfen cap.160mg, Livaro tab. 2mg

SUMMARY:
To evaluate the comparative pharmacokinetics and safety of fixed-dose combination versus coadministration of Lipilfen cap.160mg(micronized fenofibrate160mg) and Livalo tab. 2mg(pitavastatin Ca 2mg) under fed condition in healthy male volunteers.

DETAILED DESCRIPTION:
To develop combination product of micronized fenofibrate plus pitavastatin, we would like to evaluate the comparative pharmacokinetics and safety of fixed-dose combination(micronized fenofibrate160mg+pitavastatin Ca 2mg) versus coadministration of Lipilfen cap.160mg(micronized fenofibrate160mg) and Livalo tab. 2mg(pitavastatin Ca 2mg) under fed condition in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age 19 to 55 at the screening visit
* Body weight≥50kg and within Ideal body weight±20%
* Subject who is judged to be eligible according to clinical laboratory tests including hematological examination, blood chemistry examination, urine analysis
* Subject who volunteerly determined to participate in and agreed to comply with precautions after totally understand the detailed explanations about this study

Exclusion Criteria:

* Subject with serious active cardiovascular, respiratory, hepatology, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
* Subject with symptoms of acute disease within 28days prior to study medication dosing
* Subject with known for history which affect on the absorption, distribution, metabolism or excretion of drug
* Subject with clinically significant active chronic disease
* Subject with any of the following conditions in laboratory test i. AST(aspartate aminotransferase) or ALT(alanine transferase) > upper normal limit × 1.5 ii. Total bilirubin > upper normal limit × 1.5 iii. renal failure with Creatinine clearance < 50mL/min iv. creatine phosphokinase > upper normal limit × 2
* Positive test results for hepatitis B virus surface antigen, anti-hepatitis C virus antibody, human immunodeficiency virus antigen/antibody,venereal disease research laboratory test
* Use of any prescription medication within 14 days prior to study medication dosing
* Use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
* Subject with clinically significant allergic disease (except for mild allergic rhinitis and mild allergic dermatitis that are not needed to administer drug)
* Subject with known for hypersensitivity reaction to fenofibrate, fenofibric acid or statin
* gallbladder disease
* Subject who experiences photo-allergy or photo-toxicity during administrating fibrates or ketoprofen
* Subject with genetic deficiency such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
* Subject who is not able to taking the institutional standard meal
* Subject with whole blood donation within 60days, component blood donation within 20days
* Subjects receiving blood transfusion within 30days prior to study medication dosing
* Participation in any clinical investigation within 60days prior to study medication dosing
* Continued excessive use of caffeine (caffeine > five cups/day), alcohol(alcohol>30g/day) and severe heavy smoker(cigarette > 10 cigarettes per day)
* Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
AUClast(area under the curve) of fenofibric acid | Pre-dose(0h), 1, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72, 96h(15 points)
Cmax(maximum concentration) of fenofibric acid | Pre-dose(0h), 1, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72, 96h(15 points)
AUClast(area under the curve) of pitavastatin | Pitavastatin : Pre-dose(0h), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72h(18 points)
Cmax(maximum concentration) of pitavastatin | Pitavastatin : Pre-dose(0h), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72h(18 points)

SECONDARY OUTCOMES:
AUCinf(area under the curve) of fenofibric acid | Pre-dose(0h), 1, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72, 96h(15 points)
Tmax(time to Maximum Plasma Concentration) of fenofibric acid | Pre-dose(0h), 1, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72, 96h(15 points)
t1/2(half life) of fenofibric acid | Pre-dose(0h), 1, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72, 96h(15 points)
AUCinf(area under the curve) of pitavastatin | Pre-dose(0h), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72h(18 points)
Tmax(time to Maximum Plasma Concentration) of pitavastatin | Pre-dose(0h), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72h(18 points)
t1/2(half life) of pitavastatin | Pre-dose(0h), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 8, 12, 24, 48, 72h(18 points)
Number of participants with adverse events | Participants will be followed for the duration of hospital stay, and expected period for maximum 7 days from the discharge

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea